CLINICAL TRIAL: NCT02463214
Title: Prevention of Healthcare Associated Infections in Bone Marrow Transplant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health Research Institute (Other)
Responsible Party: Principal Investigator, Linda Hoang, Medical Microbiologist, BC Centre for Disease Control, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H15-00662
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Transplantation Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Room (No Intervention): Standard bone marrow transplant recovery, single occupancy, room
- Engineered Room (Experimental): Single occupancy bone marrow transplant recovery room, engineered with touchless devices, and surfaces coated with either copper or titanium dioxide.
  Interventions: Other: Engineered Room

INTERVENTIONS:
Other: Engineered Room — Touchless devices:
  Hand sanitizers, faucets, paper towel dispensers, call devices, Ultraviolet C Aseptix™ Disinfection devices above bathroom doors
  Copper products:
  Room and bathroom entrance door hardware, over bed table and bed side table surfaces, chair metal arms, wardrobe handles and knobs, weigh scale, sinks, grab bars, light switch panels, toilet flush handles, faucets and handles, patient bed rails.
  Titanium dioxide paint:
  Room walls, head walls, light switches, bathroom wall shelves, toilet tank and bowl, head wall unit fixed equipment, television remote and Bed Control remote
  Arms: Engineered Room

SUMMARY:
This study involves sampling bone marrow transplant patients, hospital workers and the patient room for microbes using swabs and other techniques. We send these samples to the laboratory, where they will use state-of-the art technology to identify and relate the microbes to each other. This study also involves putting copper, nickel, or titanium into some hospital rooms, and seeing whether these metals influences the growth of microbes. Some equipment in the hospital room, such as faucets and soap dispensers will be replaced by sensor-based (e.g. touchless) controls.

DETAILED DESCRIPTION:
Bacteria and other microbes are everywhere, the majority of which are harmless. They live on our bodies, on everyday objects, in food, and in our environment. They are passed around through the many interactions with other people and our surroundings. Some are even beneficial, helping us digest our food or protecting us from infections caused by harmful microbes.

In rare instances, some of the harmful microbes can cause infections. When a microbe causes an infection while we are in healthcare facilities, they are called "Healthcare-associated infections", or "HAIs". Examples that you may have heard of include Clostridium difficile, and MRSA (methicillin-resistant Staphylococcus aureus). Vancouver General Hospital already has some of the lowest HAI rates in the country. We have dedicated hospital workers that do a great job at preventing HAIs, but we are always looking for ways to be even better.

ELIGIBILITY:
Inclusion Criteria (Patients):

* undergoing allogenic bone marrow transplant for acute myeloid leukemia
* will be admitted to the leukemia and bone marrow transplant service at Vancouver General Hospital
* admission to the ward anticipated to be approximately 28 days

Exclusion Criteria (Patients):

* allergies to copper, nickel or titanium
* patients admitted for stays anticipated to be less than 28 days

Inclusion Criteria (Health care worker):

* undergoing allogenic bone marrow transplant for acute myeloid leukemia
* caring for patient enrolled in the study as a primary nurse

Exclusion Criteria (Health care worker):

* allergies to copper, nickel or titanium

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-09; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change in bioburden on surfaces | up to 28 days
  Looking to see the effectiveness of copper and titanium on the microbiota in the environment of the recovery room.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Hoang, MD FRCPC, Principal Investigator — The University of British Columbia; Elizabeth Bryce, MD FRCPC, Principal Investigator — The University of British Columbia; Patrick Tang, MD PhD FRCPC, Principal Investigator — Sidra Medicine
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada